CLINICAL TRIAL: NCT04672915
Title: Prevalence of Occult Hepatitis B Virus Infection（OBI） in Subjects With Chronic Hepatitis B (CHB） Family History and Cascading of Care Linked to Treatment in West China
Brief Title: Prevalence of Occult Hepatitis B Virus Infection（OBI） in Subjects With Chronic Hepatitis B（CHB） Family History
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: HX202047
Record Dates: First submitted 2020-11-18; First posted 2020-12-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-08

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: test of HBV DNA — Real time PCR or nested PCR to check

SUMMARY:
Mother to Child transmission is the main route of hepatitis B virus (HBV) transmission in China, attributing to over 50% HBV infection. Familial aggregation in HBV infection is well recognized with underlying stipulations like mother-to-child transmission（MTCT）, susceptible genes, close contact and other factors. Not surprisingly, a large proportion of hepatitis B virus infected population in China have a family history of hepatitis B virus infection. In clinical practice those family members usually undergo merely hepatitis B virus serology tests without HBV DNA test, which ruled out false HBsAg (-) or Occult HBV Infection (OBI) from Screening and linkage to care (SLTC). Unfortunately, the missed-out OBI in CHB family members was of a greater prevalence compared to those from general population (8.0% vs. 2.6%) . Moreover, OBI has been well recognized as strong risk factor in hepatocellular carcinoma （HCC） development with significant HBV DNA integration into host genome . In light of the latest 2019 China CHB guidelines, treatment criteria covered subjects with family history of CHB related cirrhosis or hepatocellular carcinoma(HCC). Therefore, subjects of HBsAg (+) with normal alanine aminotransferase（ALT） or OBI are eligible for further consideration of HBV anti-viral treatment.

This study proposed will explore the prevalence of OBI in subjects with family history of HBV related cirrhosis or HCC. The screened HBsAg (+) with normal alanine aminotransferase(ALT) and OBI subjects would be linked to anti-viral therapies.

DETAILED DESCRIPTION:
Serum samples were tested for liver enzymes and liver synthesis function including ALT, aspartate aminotransferase（AST）, and albumin, etc. using a Hitachi 7600 automatic analyzer and reagent system (Hitachi, Tokyo, japan). HBsAg quantification was performed using automated electrochemiluminescence Immunoassay (ECLIA) manufactured by Roche. HBsAb, HBeAg, HBeAb and HBcAb were measured semi-quantitatively using Chemiluminescence Immunoassay (CLIA) manufactured by Abbott Diagnostics (USA). Serum HBV DNA levels were measured using the COBAS TaqMan HBV Monitor Test, with a lower limit of detection of 20 IU/mL (100 copies/mL).

The false negative result excluding OBI due to Real time PCR (lower limit of 20 IU/ml) technically may exist. The study group plan to carry out nested PCR (specifically target the HBV Pre-S, S, Pre-C/Core, and X open reading frames) on subjects with HBsAg (-) HBV DNA (-) and HBcAb(+) to double check the potential false negative result in HBV DNA from Real time PCR. Quantitation of intrahepatic HBV cccDNA by quantitative real-time PCR (qPCR).

ELIGIBILITY:
Inclusion Criteria:

* First- and second-degree relatives of CHB patients in west China；
* Subjects with family history of CHB related cirrhosis or HCC;
* Subjects with ability to understand and sign a written informed consent form.

Exclusion Criteria:

* Positive antibody against hepatitis C virus(HCV),hepatitis D Virus(HDV), or human immunodeficiency virus(HIV) (anti-HCV, anti-HDV, or anti-HIV)
* Evidence of other autoimmune or metabolic liver diseases (except non-alcoholic fatty liver disease).
* Moribund state including advanced/pre-terminal liver cancer or other non-hepatic cancers
* Non-hepatic cancer undergoing chemotherapy within last 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population from the family with the history of CHB related cirrhosis or HCC.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of OBI in subjects with CHB family history | 1 year
  Serum samples were tested for liver enzymes and liver synthesis function including ALT, Aspartate aminotransferase（AST）, and albumin, etc. using a Hitachi 7600 automatic analyzer.HBsAg quantification was performed using automated electrochemiluminescence Immunoassay (ECLIA) manufactured by Roche, with limit of detection at 0.05 IU/mL or confirmed by the HBsAg confirmatory assay ,with limit of detection at 0.005 IU/mL. HBsAb, HBeAg, HBeAb and HBcAb were measured semi-quantitatively using Chemiluminescence Immunoassay (CLIA) manufactured by Abbott Diagnostics (USA). Serum HBV DNA levels were measured using the COBAS TaqMan HBV Monitor Test, with a lower limit of detection of 20 IU/mL (100 copies/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Yingren Zhao, Study Director — First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- First Affiliated Hospital of Xi'an JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided